CLINICAL TRIAL: NCT06299241
Title: Evaluation of Physical Performance in Old Adults With Sarcopenic Obesity
Acronym: PREFISAR
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C313
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Sarcopenia
Keywords: Aging; Obesity; Sarcopenia; Physical performance
MeSH Terms: conditions — Obesity; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objectives of the present study are to estimate the sarcopenic proportion in a cohort of obese older subjects who have been hospitalized. The secondary objective is to individuate several clinical variables that differ between the sarcopenic obese patient and the not sarcopenic obese patient.

DETAILED DESCRIPTION:
80 obese patients of both genders (BMI > 35), with an age > 60 years, hospitalized at the Hospital San Giuseppe, Istituto Auxologico Italiano, IRCCS, Piancavallo (VB) are selected. For each patient, the following information are collected at the time of admission:

* anthropometric parameters (height, weight, BMI, waist and hip circumference);
* body composition (free fat mass, fat mass), measured with impedance (BIA) and DEXA;
* hand strength measured with the hand grip test;
* explosive strength of lower limbs, measured with the stair climbing test;
* Senior Fitness Test (SFT), a battery of tests useful to estimate the fitness level in the elderly. SFT is a test that leads to measuring different physical parameters typical of daily activities: strength of upper and lower limbs, aerobic resistance, flexibility of lower and upper limbs, agility, and dynamic equilibrium. The measurements obtained make it possible to classify the skills as high function or low function.
* Physical performance test (PPT), which evaluates 7 physical capabilities areas of the subject to perform actions during daily life. The cut-off to determine the motor limitation condition is a score of ≤ 20 (out of 28 points).
* Questionnaire SF-12 (Short Form Health Survey), which leads to a multi-dimensional measuring of the life quality related to health. It is composed of 12 questions from which can be obtained two synthetic indices, one related to physical health and one related to mental health.
* Oswestry Disability Index questionnaire, elaborated to have information on how back problems, or leg problems, can influence physical abilities related to daily life.

The presence of sarcopenia is identified based on the European Working Group on Sarcopenia in Older People (EWGSOP2) (Cruz-Jentoft AJ et al. 2019) definition. The physical performance parameters is evaluated according to the age, sex, obesity grade, and presence of sarcopenic obesity.

ELIGIBILITY:
Inclusion Criteria:

* obese patients (BMI > 35),
* both genders
* age > 60 years
* hospitalization at San Giuseppe Hospital, Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), Italy for a multidisciplinary 3-week body weight reduction program

Exclusion Criteria:

* obese patients with BMI < 35
* age < 60 years

Ages: 60 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Obese patients (BMI > 35), of both genders, aged > 60 years, hospitalized at San Giuseppe Hospital, Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), Italy for a multidisciplinary 3-week body weight reduction program.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Fat free mass | Baseline
  Measurement of body composition parameters with bioimpedance analysis (BIA) and DEXA
Evaluation of lower limb muscle strength | Baseline
  Measurement with the stair climbing test
Senior Fitness Test (SFT) | Baseline
  A battery of tests useful to estimate the fitness level of the elderly. This is a test that allows measuring different physical parameters typical of daily activities: strength of upper and lower limbs, aerobic resistance, flexibility of lower and upper limbs, agility, and dynamic equilibrium.
Physical performance test (PPT) | Baseline
  A test evaluating 7 physical capabilities areas of the subject to perform actions during daily life. The cut-off to determine the motor limitation condition is a score of ≤ 20 (out of 28 points).
Fat mass | Baseline
  Measurement of body composition parameters with bioimpedance analysis (BIA) and DEXA;

SECONDARY OUTCOMES:
Questionnaire SF-12 (Short Form Health Survey) | Baseline
  A questionnaire allowing a multi-dimensional measurement of quality of life related to health. It is composed of 12 questions from which it is possible obtaining two synthetic indexes, one related to physical health and the other one related to mental health.
Oswestry Disability Index questionnaire | Baseline
  A questionnaire elaborated to have information on how back problems, or leg problems, can influence physical abilities related to daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Site Piancavallo, Oggebbio, Verbania, Italy